CLINICAL TRIAL: NCT00646191
Title: Multicenter Extension Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello / Director, Clinical Program Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-529
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: adalimumab
- B (Active Comparator)
  Interventions: Drug: adalimumab
- C (Active Comparator)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — 40 mg eow through Week 12 followed by OL 40 mg eow through Week 48, permitted to escalate to weekly dosing upon relapse
  Other Names: ABT-D2E7; Humira
  Arms: A
Drug: adalimumab — 40 mg weekly through Week 48 (OL Week 12 - 48)
  Other Names: ABT-D2E7; Humira
  Arms: B
Drug: adalimumab — 80 mg W0, 40 mg eow through Week 12 followed by OL 40 mg eow through Week 48, permitted to escalate to weekly dosing upon relapse
  Other Names: ABT-D2E7; Humira
  Arms: C

SUMMARY:
Study of the Safety and Efficacy of Adalimumab in Subjects with Moderate to Severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject completed prior PS study

Exclusion Criteria:

* Subject has other active skin diseases
* Multiple concomitant therapy restrictions and/or washouts (topicals, UV, other systemic PS therapies)
* Poorly controlled medical conditions
* History of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease
* History of cancer or lymphoproliferative disease
* History of active TB or listeriosis, or persistent chronic or active infections
* Known to have immune deficiency or is immunocompromised
* Clinically significant abnormal laboratory test results
* Erythrodermic psoriasis or generalized pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2003-03; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | Week 12
Adverse Events | Throughout Study Participation

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index | Week 0, 4, 8, 12, 16, 20, 24, 32, 40 and 48
DLQI, SF-36, Zung Depression Self-Rating Scale, EQ-5D, VAS | Week 12, 24 and 48
Physician's Global Assessment | Week 12, 16, 20, 24, 32, 40 and 48